CLINICAL TRIAL: NCT01769209
Title: A Phase II Study of Subcutaneous Bortezomib in Combination With Chemotherapy (VXLD) for Relapsed/Refractory Adult Acute Lymphoblastic Leukemia
Brief Title: Bortezomib and Combination Chemotherapy in Treating Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Michaela Liedtke, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-25596; NCI-2012-03094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HEMALL0008 (Other: OnCore Number); IRB-25596 (Other: Stanford IRB)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2018-10-09 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: B-cell Adult Acute Lymphoblastic Leukemia (ALL); Ph-positive Adult Acute Lymphoblastic Leukemia (ALL); Recurrent Adult Acute Lymphoblastic Leukemia (ALL); T-cell Adult Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Bortezomib; Doxorubicin; pegaspargase; Vincristine; Dexamethasone; Calcium Dobesilate; Cytarabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bortezomib + Chemotherapy (Experimental): Patients receive bortezomib on Days 1, 4, 8, and 11; doxorubicin hydrochloride on Day 1; PEG-asparaginase on Days 5 and 22; vincristine sulfate on Days 1, 8, 15, and 22; dexamethasone daily on Days 1 to 14; cytarabine on Day 1, and methotrexate on Day 15.
  Interventions: Drug: Bortezomib; Drug: Doxorubicin hydrochloride (HCl); Drug: PEG-Asparaginase; Drug: Vincristine sulfate; Drug: Dexamethasone; Drug: Cytarabine; Drug: Methotrexate

INTERVENTIONS:
Drug: Bortezomib — Administered subcutaneously (SC) at 1.3 mg/m², on Days 1, 4, 8, and 11.
  Other Names: Velcade; LDP 341; MLN341
Drug: Doxorubicin hydrochloride (HCl) — Administered intravenously (IV) over 15 min at 60mg/m², on Day 1.
  Other Names: Adriamycin; Adriamycin PFS; Adriamycin RDF; Adria; ADM; ADR; Rubex; VXLD
Drug: PEG-Asparaginase — Administered intravenously (IV) or intramuscularly (IM) 2500 U/m² (maximum 3750 U), on Days 5 and 22.
  Other Names: Pegaspargase; Oncaspar; L-asparaginase with polyethylene glycol; Pegasparaginase; PEG-L-asparaginase; PEG-ASP
Drug: Vincristine sulfate — Administered by intravenous (IV) push at 1.5 mg/m² (maximum 2 mg), on Days 1, 8, 15, and 22.
  Other Names: Leurocristine sulfate; Vincasar PFS; VCR
Drug: Dexamethasone — Administered orally (PO) at 10 mg/m², daily on Days 1 to 14.
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: Cytarabine — Administered intrathecally (IT) at 100 mg, on Day 1
  Other Names: Cytosine arabinoside; ARA-C; Arabinofuranosylcytosine; Arabinosylcytosine; Cytosar-U
Drug: Methotrexate — Administered intrathecally (IT) at 15 mg, on Day 15.
  Other Names: Amethopterin; MTX

SUMMARY:
This study evaluates the value of bortezomib in combination with specified chemotherapies for the treatment of patients with relapsed or refractory acute lymphoblastic leukemia. Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

Determine the response rate of bortezomib in combination with a chemotherapy backbone of doxorubicin (doxorubicin hydrochloride), vincristine (vincristine sulfate), PEG-asparaginase (pegaspargase), and dexamethasone in patients with relapsed/refractory acute lymphoblastic leukemia.

SECONDARY OBJECTIVES:

* Estimate the rate of complete response (CR) and CR with incomplete platelet recovery (CRp) on Day 29 after re-induction.
* Determine progression-free survival (PFS) at 2 years after re-induction.
* Determine failure-free survival (FFS) at 1 year after re-induction.
* Overall survival (OS) at 1 year after re-induction.
* Assess safety and tolerability of the study drug.
* Determine whether bortezomib induces reactive oxygen species (ROS) in circulating acute lymphoblastic leukemia (ALL) blast cells.

OUTLINE:

Patients receive bortezomib subcutaneously (SC) on Days 1, 4, 8, and 11; doxorubicin hydrochloride intravenously (IV) on day 1; pegaspargase IV or intramuscularly (IM) on Days 5 and 22; vincristine sulfate IV on days 1, 8, 15, and 22; dexamethasone orally (PO) daily on Days 1 to 14; cytarabine intrathecally (IT) on Day 1 and methotrexate intrathecally (IT) on Day 15. Patients with central nervous system disease receive intrathecal treatment per investigator's discretion.

Participants are followed up every 3 months for up to 2 years after completion of study treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Voluntary written informed consent
* Female subjects who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 30 days after the last dose of bortezomib, or agree to completely abstain from heterosexual intercourse
* Male subjects, even if surgically sterilized (ie, status post vasectomy) who:

  * Agree to practice effective barrier contraception during the entire study treatment period and through a minimum of 30 days after the last dose of study drug, OR
  * Agree to completely abstain from heterosexual intercourse
* • Relapsed or refractory B or T cell acute lymphoblastic leukemia that has progressed following at least one prior therapy. Ph+ patients are eligible. Relapsed ALL is defined in patients as the reappearance of leukemia cells in the peripheral blood or bone marrow or appearance of extramedullary disease after a complete remission. Refractory ALL is defined in patients as failure to achieve a complete remission after induction therapy. Complete remission is defined by <5% leukemia cells in the bone marrow with recovery of peripheral blood counts. Relapsed disease can be documented by bone marrow biopsy (>5% cells in the bone marrow) or by flow cytometry in the peripheral blood or biopsy of extramedullary disease.
* Has received at least 1 line of prior systemic therapy that may NOT have included bortezomib (Velcade); patients who have undergone autologous/allogeneic stem cell transplantation are eligible
* Transplant-eligible patients are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* No poorly-controlled intercurrent illness including, but not limited to, ongoing or active infection, poorly controlled diabetes, symptomatic congestive heart failure, or psychiatric illness that in the opinion of the investigator would limit compliance with study requirements
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 x upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 x (ULN unless elevation is deemed due to leukemia infiltration)
* Adequate renal function defined as creatinine clearance of ≥ 30 mL/minute by the Cockcroft-Gault method

EXCLUSION CRITERIA

* > 1.5 x ULN total bilirubin
* ≥ Grade 2 peripheral neuropathy
* Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities; prior to study entry, any electrocardiogram (ECG) abnormality at screening must be documented by the investigator as not medically relevant
* Hypersensitivity to bortezomib, boron, or mannitol
* Pregnant or lactating
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study
* Diagnosed or treated for another malignancy within 2 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy
* Participation in clinical trials with other investigational agents not included in this trial throughout the duration of this trial
* Radiation therapy within 3 weeks before randomization; enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy
* Prior exposure ≥ 350 mg/m² of anthracycline (doxorubicin equivalent)
* Left ventricular ejection fraction < 40%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-11-25 (Actual); Study Completion 2017-07-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Liedtke, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bortezomib + Chemotherapy
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 37.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (RR)
Description: Response Rate (RR) was determined as the sum of complete response (CR) and partial response (PR). Due to overlap, "complete response rate without platelet recovery" (CRp) is not included in Response Rate (RR). The outcome is reported as the total number without dispersion.
  * CR = No circulating blasts or extramedullary disease; trilineage hematopoiesis; absolute neutrophil count (ANC) > 1,000/microliter; platelets > 100,000/microliter; < 5% blasts in bone marrow.
  * CRp = Meets all criteria for CR except platelet count.
  * PR = Meets all criteria for CR except bone marrow contains 5 to 25% leukemia cells.
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Participants | 11

2. Secondary Outcome: Complete Response (CR)
Description: Complete response (CR) was determined the number of participants who achieved CR by Day 29 after induction treatment. The outcome is reported as the total number without dispersion. CR is defined as:
  * CR = No circulating blasts or extramedullary disease; trilineage hematopoiesis; absolute neutrophil count (ANC) > 1,000/microliter; platelets > 100,000/microliter; < 5% blasts in bone marrow.
  * Not CR = All statuses and conditions if less than or not as defined.
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Participants | 11

3. Secondary Outcome: Complete Response Without Platelet Recovery (CRp)
Description: Complete response without platelet recovery (CR) was determined as the number of participants who achieved CRp by Day 29 after induction treatment. The outcome is reported as the total number without dispersion. The outcome reflects only those subjects that meet all complete response (CR) criteria except platelet count; participants that meet all criteria including platelet count are not included in this outcome. CR and CRp are defined below.
  * CR =.No circulating blasts or extramedullary disease; trilineage hematopoiesis; absolute neutrophil count (ANC) > 1,000/microliter; platelets > 100,000/microliter; < 5% blasts in bone marrow.
  * CRp = Meets all criteria for CR except platelet count.
Time Frame: Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Participants | 1

4. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival (PFS) was assessed as survival without progression at 2 years. The outcome is reported as the number (without dispersion) of the participants alive without progression.
  Progression = More than 25% increase in circulating and/or bone marrow blasts, or the development of extramedullary disease.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Participants | 3

5. Secondary Outcome: Failure-free Survival (FFS)
Description: Failure-free survival (FFS) was assessed as survival without progression or the addition of another systemic therapy, at or within 2 years. The outcome is reported as the number (without dispersion) of the participants alive without progression. Progression is defined below.
  Progression = More than 25% increase in circulating and/or bone marrow blasts, or the development of extramedullary disease.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Participants | 3

6. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was assessed as participants remaining alive 2 years after induction therapy. The outcome is reported as the number of participants (without dispersion).
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Participants | 5

7. Secondary Outcome: Related Adverse Events (Grade 3, 4, 5)
Description: Toxicity was assessed as related grade 3, 4, or 5 adverse events (AEs) per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03. The outcome is reported as the total numbers of events (without dispersion) by CTCAE Body System, and whether the event was a hematologic toxicity or non-hematologic toxicity.
Time Frame: 45 days
Population: Events specifically defined per protocol as "Hematologic Toxicity" or"Non-hematologic Toxicity" are included under the specific Body System and as a Hematologic or Non-hematologic Toxicity.
Measure: Number; unit: Treatment-related adverse events
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 18
Treatment-related adverse events
  Blood and Lymphatic System Disorders | 109
  Gastrointestinal Disorders | 9
  Hepatobiliary disorders | 2
  Infections and Infestations | 17
  Investigations | 78
  Metabolism and Nutrition Disorders | 49
  Nervous System Disorders | 1
  Respiratory, Thoracic and Mediastinal Disorders | 1
  Vascular Disorders | 2
  Hematologic Toxicity | 63
  Non-hematologic Toxicity | 52

8. Secondary Outcome: Induction of Reactive Oxygen Species (ROS)
Description: Circulating acute lymphoblastic leukemia (ALL) blast cells were to be evaluated for the presence of reactive oxygen species (ROS).
Time Frame: 2 years
Population: Assay development was unsuccessful, and the assessment and analysis were not conducted for any samples.
Arm/Group | Bortezomib + Chemotherapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Bortezomib + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 13/18
Serious Adverse Events (participants affected / at risk) | 10/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib + Chemotherapy (N=18)
Neutropenic fever (febrile neutropenia) (Blood and lymphatic system disorders) | 1 (1)
Disseminated intravascular coagulation (DIC) (Blood and lymphatic system disorders) | 1 (1)
Colon and caecum inflammation (typhilitis, colitis) (Gastrointestinal disorders) | 1 (1)
Hepatobilliary Disorders-Other, veno-occlusive disease (Hepatobiliary disorders) | 1 (1)
Septic shock (sepsis) (Infections and infestations) | 5 (5)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib + Chemotherapy (N=18)
Neutropenic fever (febrile neutropenia) (Blood and lymphatic system disorders) | 5 (5)
Neutropenia (Blood and lymphatic system disorders) | 13 (13)
Lymphopenia (Blood and lymphatic system disorders) | 13 (13)
Anemia (Blood and lymphatic system disorders) | 16 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (12)
Heart palpitations (tachycardia) (Cardiac disorders) | 3 (3)
Heart failure (congestive heart failure) (Cardiac disorders) | 2 (2)
Decreased hearing (hearing impaired) (Ear and labyrinth disorders) | 1 (1)
Blurred vision (Eye disorders) | 3 (3)
Dry eyes (Eye disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Vomiting (nausea) (Gastrointestinal disorders) | 13 (13)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (7)
Gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 6 (6)
Colon and caecum inflammation (typhilitis, colitis) (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 10 (10)
Perianal pain ( Anal pain) (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2)
Swelling (edema) (General disorders) | 9 (9)
Fatigue (General disorders) | 7 (7)
Chills (General disorders) | 2 (2)
Hepatobilliary Disorders-Other, liver abscess (Hepatobiliary disorders) | 1 (1)
Infections and infestations-Other,thrush (Infections and infestations) | 3 (3)
Respiratory infections (Infections and infestations) | 8 (8)
Infections and infestations-Other, Herpes simplex virus (Infections and infestations) | 2 (2)
Septic shock (sepsis) (Infections and infestations) | 1 (1)
Respiratory syncytial virus (RSV) (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 3 (3)
Infections and infestations-Other, Herpes simplex virus Line, sepsis (Infections and infestations) | 5 (5)
Fibrinogen decreased (Investigations) | 17 (17)
Partial thromboplastin time (PTT) high (Investigations) | 7 (7)
Aspartate aminotransferase (AST) elevated (Investigations) | 14 (14)
Alanine aminotransferase (ALT) elevated (Investigations) | 15 (15)
Bilirubin elevated (Investigations) | 11 (11)
Alkaline Phosphatase elevated (Investigations) | 9 (9)
Gamma-glutamyl transferase (GGT) elevated (Investigations) | 2 (2)
Amylase high (Investigations) | 3 (3)
Lipase high (Investigations) | 6 (6)
Creatinine high (Investigations) | 7 (7)
Apetite loss (anorexia) (Metabolism and nutrition disorders) | 5 (5)
Hypoalbuminemia (Albumin low) (Metabolism and nutrition disorders) | 18 (18)
Hypertriglyceridemia (Triglycerides high) (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia -Sodium high (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia -Sodium low (Metabolism and nutrition disorders) | 5 (5)
Hypokalemia -Potassium low (Metabolism and nutrition disorders) | 12 (12)
Hyperkalemia -Potassium high (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesemia -Magnesium low (Metabolism and nutrition disorders) | 9 (9)
Hypocalcemia -Calcium low (Metabolism and nutrition disorders) | 13 (13)
Hypophosphatemia -Phosphorus low (Metabolism and nutrition disorders) | 9 (9)
Metabolism and Nutrition Disorders-Other Phosphorus high (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Glucose high) (Metabolism and nutrition disorders) | 13 (13)
Hypoglycemia -Glucose low (Metabolism and nutrition disorders) | 3 (3)
Leg weakness (generalized muscle weakness ) (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 13 (13)
Avascular necrosis (Bone infarct) (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 3 (3)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8)
Seizures (Nervous system disorders) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Restless leg (akathisia) (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 13 (13)
Intracranial hemorrhage (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pain during urination (dysuria) (Renal and urinary disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Breath shortness (Dyspnea) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest pain (pleuritic pain) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nosebleed (Epistaxis) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration -Lip lesion (Skin and subcutaneous tissue disorders) | 1 (1)
High blood pressure (hypertension) (Vascular disorders) | 2 (2)
Low blood pressure (hyportension) (Vascular disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No